CLINICAL TRIAL: NCT01482884
Title: A Phase IIa, Randomised, Double-blind, Placebo-controlled, Parallel-arm, Multicenter Study to Evaluate the Efficacy and Safety of Tralokinumab (CAT-354), a Recombinant Human Monoclonal Antibody Directed Against Interleukin-13 (IL-13), as add-on Therapy, on Clinical Response in Patients With Active, Moderate-to-severe, Ulcerative Colitis
Brief Title: Evaluation of Efficacy and Safety of Tralokinumab in Patients With Active, Moderate-to-severe Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: MedImmune Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D2211C00001; EudraCT number 2011-004812-40
Record Dates: First submitted 2011-11-29; First posted 2011-12-01 (Estimated); Results first posted 2016-04-05 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-03

CONDITIONS: Ulcerative Colitis
Keywords: tralokinumab; inflammatory bowel disease; moderate to severe ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — tralokinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): tralokinumab (CAT-354) sc injection
  Interventions: Drug: tralokinumab
- 2 (Placebo Comparator): placebo sc injection
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: tralokinumab — 2 sc injections of every 2 weeks for 12 weeks.
  Arms: 1
Drug: placebo — 2 sc injections of every 2 weeks for 12 weeks.
  Arms: 2

SUMMARY:
The study is designed to evaluate the clinical efficacy and safety of tralokinumab as compared to placebo. Investigational product will be administered as subcutaneous injection. All patients will continue background therapy for ulcerative colitis as per local standards of care in addition to investigational product.

DETAILED DESCRIPTION:
A phase IIa, randomised, double-blind, placebo-controlled, parallel-arm, multicenter study to evaluate the efficacy and safety of tralokinumab (CAT-354), a recombinant human monoclonal antibody directed against interleukin-13 (IL-13), as add-on therapy, on clinical response in patients with active, moderate-to-severe, ulcerative colitis

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed ulcerative colitis at least 90 days prior randomisation.
* Men or women age 18 - 75 years.
* Non-hospitalized patients with moderate-severe ulcerative colitis treated with stable background UC therapy (e.g. containing 5-aminosalicylates, and/or low dose of glucocorticosteroids, and/or purine analogue) prior to randomization.
* Females of childbearing potential who are sexually active with a nonsterilized male partner must use highly effective contraception from Day1.
* Nonsterilized males or sterilized males who are ≤1 year post-vasectomy who are sexually active with a female partner of childbearing potential must use a highly effective method of contraception.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* History of colostomy.
* Current diagnosis of indeterminate colitis, Crohn's disease, ischemic colitis, fulminant colitis and/or toxic megacolon and patients with ulcerative colitis limited to the rectum (ulcerative proctitis).
* Hepatitis B, C or HIV.
* History of cancer.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Berner Hansen, MD, PhD, Study Director — AstraZeneca R&D Mölndal Pepparedsleden 1, S-431 83 Mölndal, Sweden; Silvio Danese, MD, PhD, Principal Investigator — IBD Center, Instituto Clinico Humanitas, Department of Gastroenterology, Via Manzoni 56, 20089 Rozzano, Milan, Italy
Locations (28):
- Czechia (4):
  - Research Site, České Budějovice
  - Research Site, Hradec Králové
  - Research Site, Olomouc
  - Research Site, Prague
- France (7):
  - Research Site, Amiens
  - Research Site, Caen
  - Research Site, Clichy
  - Research Site, Nice
  - Research Site, Pessac
  - Research Site, Rouen
  - Research Site, Vandœuvre-lès-Nancy
- Germany (4):
  - Research Site, Ludwigshafen
  - Research Site, Oelde
  - Research Site, Potsdam
  - Research Site, Wangen
- Italy (4):
  - Research Site, Florence
  - Research Site, Padua
  - Research Site, Roma
  - Research Site, Rozzano
- Poland (5):
  - Research Site, Bydgoszcz
  - Research Site, Częstochowa
  - Research Site, Lodz
  - Research Site, Sopot
  - Research Site, Warsaw
- United Kingdom (4):
  - Research Site, Cambridge
  - Research Site, Coventry
  - Research Site, Oxford
  - Research Site, Shrewsbury

REFERENCES:
- [Result] Danese S, Rudzinski J, Brandt W, Dupas JL, Peyrin-Biroulet L, Bouhnik Y, Kleczkowski D, Uebel P, Lukas M, Knutsson M, Erlandsson F, Hansen MB, Keshav S. Tralokinumab for moderate-to-severe UC: a randomised, double-blind, placebo-controlled, phase IIa study. Gut. 2015 Feb;64(2):243-9. doi: 10.1136/gutjnl-2014-308004. Epub 2014 Oct 10. PMID 25304132
- See also: D2211C00001_Protocol_Redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1241&filename=D2211C00001_Protocol_Redacted.pdf
- See also: D2211C00001_Study_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1241&filename=D2211C00001_Study_Synopsis_with_changes.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 147/111 patients were enrolled/randomized from 31 centres in 6 European countries. The first patient was enrolled on 26 March 2012, and the last patient completed the study on 24 June 2013.
Pre-assignment Details: Participants were enrolled for a period of 3 weeks.
Groups:
- Tralokinumab: Tralokinumab 300 mg was administered during study as two subcutaneous 150 mg injections every 2 weeks for 12 weeks starting from Visit 2.
- Placebo: Placebo was administered during study as two subcutaneous injections every 2 weeks for 12 weeks starting from Visit 2.
Period: Overall Study
Arm/Group | Tralokinumab | Placebo
Started | 56 (One participant did not receive study treatment) | 55
Completed | 43 | 37
Not Completed | 13 | 18
Not completed — Medical decision due to lack of efficacy | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 2 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 8 | 13

BASELINE CHARACTERISTICS:
Population: All randomised participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tralokinumab | Placebo | Total
Number analyzed (Participants) | 56 | 55 | 111
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.2 (11.54) | 40.8 (13.26) | 41.5 (12.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 29 | 58
  Male | 27 | 26 | 53
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 2 | 0 | 2
  White | 54 | 54 | 108
  Other | 0 | 1 | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Asian (Other than Chinese And Japanese) | 2 | 0 | 2
  Not Applicable | 35 | 40 | 75
  Other | 17 | 13 | 30
Duration of disease [Mean (Standard Deviation); unit: Years] | 9.22 (8.523) | 7.78 (8.664) | 8.51 (8.585)
Mayo score at baseline [Mean (Full Range); unit: Scores on scale] — Mayo score is the sum of four sub-scores: stool frequency, rectal bleeding, endoscopy findings and the physician's global assessment. The total Mayo score ranges from 0-12, with higher scores indicating a more severe disease.
  Scores on scale | 8.36 [5.0 to 11.0] | 8.33 [6.0 to 11.0] | 8.34 [5.0 to 11.0]
Partial Mayo score at baseline [Mean (Full Range); unit: Scores on scale] — The partial Mayo score is the sum of the three sub-score areas: stool frequency, rectal bleeding, and the physician's global assessment.The partial Mayo score ranges from 0-9, with higher scores indicating a more severe disease.
  Scores on scale | 5.91 [3.0 to 8.0] | 5.85 [3.0 to 8.0] | 5.88 [3.0 to 8.0]
Glucocorticosteroid-refractory status [Number; unit: Participants] — Yes: if participants had received a glucocorticosteroid treatment prior to baseline and the outcome of that treatment was no improvement. No: If the outcome of the treatment was improvement or missing. Unknown: If the outcome of the treatment was unknown.
  Participants
    Yes | 3 | 8 | 11
    No | 53 | 46 | 99
    Unknown | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response at Week 8 Based on Mayo Score
Description: Clinical response was measured as a decrease in Mayo score of ≥3 points from baseline, decrease in the total Mayo score from baseline ≥30 percentage and a decrease in the sub score for rectal bleeding ≥1 or absolute sub score for rectal bleeding of 0 or 1 point. Mayo score is sum of four sub-scores: stool frequency, rectal bleeding, endoscopy findings and the physician's global assessment. The total Mayo score ranges from 0-12, with higher scores indicating a more severe disease.
Time Frame: Eight week treatment period
Population: The full analysis set consist of all randomised participants
Measure: Number; unit: Percentage of responders
Arm/Group | Tralokinumab | Placebo
Number analyzed (Participants) | 56 | 55
Percentage of responders | 37.5 | 32.7
Statistical Analysis 1: Comparison: Tralokinumab vs Placebo; The null hypothesis is that the proportion of participants responding on tralokinumab is less than or equal to the proportion of participants responding on placebo; Test type: Superiority or Other; p = 0.4062, Cochran-Mantel-Haenszel — Glucocorticosteroid-refractory status as stratification factor; Risk Difference (RD) = 4.8, 95% CI 2-sided [-13.0 to 22.5]

2. Secondary Outcome: Change in Mayo Score From Baseline to Week 8
Description: Mayo score is sum of four sub-scores: stool frequency, rectal bleeding, endoscopy findings and the physician's global assessment. The total Mayo score ranges from 0-12, with higher scores indicating a more severe disease. Change from baseline: Mayo score at week 8 minus the Mayo score at baseline.
Time Frame: Eight week treatment period
Population: The full analysis set consist of all randomised participants however the numbers for the endpoints mentioned for this secondary outcome are lower due to missing data.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Tralokinumab | Placebo
Number analyzed (Participants) | 45 | 42
Score on scale | -2.41 (0.58) | -1.92 (0.56)
Statistical Analysis 1: Comparison: Tralokinumab vs Placebo; Test type: Superiority or Other; p = 0.3937, ANCOVA; Mayo score at baseline as a covariate, and treatment and glucocorticosteroid-refractory status as factors in the model; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-1.63 to 0.65], Standard Error of Mean 0.57

3. Secondary Outcome: Mucosal Healing at Week 8 Based on Mayo Score
Description: Improvement of the endoscopy sub score (from the Mayo score) from 3 or 2 to 0 or 1 point, or from 1 to 0 points.
Time Frame: Eight week treatment period
Population: The full analysis set consist of all randomised participants
Measure: Number; unit: Percentage of participants
Arm/Group | Tralokinumab | Placebo
Number analyzed (Participants) | 56 | 55
Percentage of participants | 32.1 | 20.0
Statistical Analysis 1: Comparison: Tralokinumab vs Placebo; Test type: Superiority or Other; p = 0.1043, Cochran-Mantel-Haenszel — Glucocorticosteroid-refractory status as stratification factor; Risk Difference (RD) = 12.1, 95% CI 2-sided [-4.0 to 28.3]

4. Secondary Outcome: Clinical Remission at Week 8 Based on Mayo Score
Description: Participants were classified as in remission if Mayo score of ≤2 with no individual sub score exceeding 1 point. Mayo score is sum of four sub-scores: stool frequency, rectal bleeding, endoscopy findings and the physician's global assessment. The total Mayo score ranges from 0-12, with higher scores indicating a more severe disease.
Time Frame: Eight week treatment period
Population: The full analysis set consist of all randomised participants
Measure: Number; unit: Percentage of participants
Arm/Group | Tralokinumab | Placebo
Number analyzed (Participants) | 56 | 55
Percentage of participants | 17.9 | 5.5
Statistical Analysis 1: Comparison: Tralokinumab vs Placebo; Test type: Superiority or Other; p = 0.0326, Cochran-Mantel-Haenszel — Glucocorticosteroid-refractory status as stratification factor; Risk Difference (RD) = 12.4, 95% CI 2-sided [0.7 to 24.1]

5. Secondary Outcome: Change From Baseline in Partial Mayo Score
Description: The partial Mayo score is the sum of the three sub-score areas: stool frequency, rectal bleeding, and the physician's global assessment.The partial Mayo score ranges from 0-9, with higher scores indicating a more severe disease. Change from baseline: Mayo score at each post-baseline timepoint (week 4, 8, 12, 16, 20, and 24) minus the Mayo score at baseline.
Time Frame: From baseline to Week 4, 8, 12, 16, 20, and 24.
Population: The full analysis set consist of all randomised participants
Measure: Mean (Full Range); unit: Score on scale
Arm/Group | Tralokinumab | Placebo
Number analyzed (Participants) | 56 | 55
Score on scale
  Week 4 | -1.8 (0.31) [-8 to 3] | -0.8 (0.31) [-6 to 4]
  Week 8 | -2.4 (0.29) [-6 to 3] | -1.7 (0.30) [-6 to 1]
  Week 12 | -2.7 (0.34) [-7 to 3] | -2.6 (0.36) [-8 to 4]
  Week 16 | -2.6 (0.34) [-7 to 3] | -3.3 (0.37) [-7 to 2]
  Week 20 | -3.0 (0.33) [-7 to 2] | -3.6 (0.37) [-8 to 1]
  Week 24 | -3.0 (0.35) [-7 to 3] | -3.6 (0.38) [-7 to 1]

6. Secondary Outcome: Change From Baseline in Modified Riley Score
Description: Modified Riley score is biopsy grade which range from 0-5; where 0: Normal mucosa, 1: Infiltration of lymphocytes and plasma cells in the lamina propria, 2: Infiltration of neutrophils and eosinophils in the lamina propria, 3: Infiltration of neutrophils in the epithelium, 4: Crypt destruction, 5: Erosion and/or ulceration.
Time Frame: Eight week treatment period
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Grade on scale
Arm/Group | Tralokinumab | Placebo
Number analyzed (Participants) | 37 | 35
Grade on scale | -0.49 (0.23) | -0.74 (0.24)
Statistical Analysis 1: Comparison: Tralokinumab vs Placebo; Test type: Superiority or Other; p = 0.4490, ANCOVA; Modified Riley score at baseline as a covariate, and treatment as factors in the model; Mean Difference (Final Values) = 0.25, 95% CI 2-sided [-0.41 to 0.91], Standard Error of Mean 0.33

7. Secondary Outcome: Change From Baseline in C - Reactive Protein
Time Frame: From baseline to Week 4, 8, 12, 16, 20, and 24.
Population: The full analysis set consist of all randomised participants
Measure: Mean (Full Range); unit: mg/L
Arm/Group | Tralokinumab | Placebo
Number analyzed (Participants) | 56 | 55
mg/L
  Week 4 | -2.755 (0.31) [-33.00 to 25.00] | 0.510 (0.31) [-12.00 to 32.00]
  Week 8 | -1.089 (0.29) [-29.00 to 29.00] | 0.637 (0.30) [-43.00 to 46.00]
  Week 12 | -2.795 (0.34) [-46.00 to 63.00] | -1.974 (0.36) [-61.00 to 43.00]
  Week 16 | -3.490 (0.34) [-53.00 to 19.00] | 0.638 (0.37) [-61.00 to 97.00]
  Week 20 | -4.094 (0.33) [-52.00 to 43.00] | -1.467 (0.37) [-62.00 to 31.00]
  Week 24 | -2.754 (0.35) [-36.00 to 25.00] | -1.915 (0.38) [-59.00 to 36.00]

8. Secondary Outcome: Change From Baseline in Albumin
Time Frame: From baseline to Week 4, 8, 12, 16, 20, and 24.
Population: The full analysis set consist of all randomised participants
Measure: Mean (Full Range); unit: g/L
Arm/Group | Tralokinumab | Placebo
Number analyzed (Participants) | 56 | 55
g/L
  Week 4 | 0.0 (0.31) [-8 to 5] | -0.7 (0.31) [-7 to 6]
  Week 8 | 0.8 (0.29) [-7 to 8] | -0.2 (0.30) [-8 to 5]
  Week 12 | 0.3 (0.34) [-9 to 5] | -0.4 (0.36) [-8 to 5]
  Week 16 | 0.5 (0.34) [-10 to 12] | 0.4 (0.37) [-7 to 7]
  Week 20 | 1.1 (0.33) [-4 to 7] | 0.1 (0.37) [-6 to 9]
  Week 24 | 1.2 (0.35) [-4 to 8] | 0.2 (0.38) [-6 to 8]

9. Secondary Outcome: Change From Baseline in Calprotectin
Time Frame: From baseline to Week 4, 8, 12, 16, 20, and 24.
Population: The full analysis set consist of all randomised participants
Measure: Mean (Full Range); unit: ug/g
Arm/Group | Tralokinumab | Placebo
Number analyzed (Participants) | 56 | 55
ug/g
  Week 4 | 69.45 (0.31) [-1068.0 to 931.0] | 198.80 (0.31) [-1315.0 to 4188.0]
  Week 8 | 86.47 (0.29) [-894.2 to 912.0] | -250.52 (0.30) [-4005.0 to 4505.0]
  Week 12 | -39.19 (0.34) [-1109.0 to 841.0] | 50.31 (0.36) [-1234.0 to 4811.0]
  Week 16 | -75.10 (0.34) [-1008.0 to 1056.0] | -338.76 (0.37) [-3857.0 to 1138.0]
  Week 20 | 32.55 (0.33) [-1155.0 to 4669.0] | -402.81 (0.37) [-3835.0 to 794.0]
  Week 24 | -136.78 (0.35) [-1120.0 to 617.0] | -267.58 (0.38) [-1172.0 to 824.0]

10. Secondary Outcome: Serum Concentration of Tralokinumab
Time Frame: Pre-dose sampling at baseline, Week 4, 8, 12, 16, 20, and 24.
Population: The safety analysis set consist of all randomised participants who received at least one dose of study medication.
Measure: Mean (Full Range); unit: ug/ml
Arm/Group | Tralokinumab | Placebo
Number analyzed (Participants) | 55 | 55
ug/ml
  pre-dose at baseline | 0.00 (0.31) [0.000 to 0.000] | NA [NA to NA] — Not calculable because below the lower limit of quantification
  Week 4 | 37.9 (0.29) [12.2 to 92.2] | NA [NA to NA] — Not calculable because below the lower limit of quantification
  Week 8 | 50.2 (0.34) [5.83 to 116] | NA [NA to NA] — Not calculable because below the lower limit of quantification
  Week 12 | 48.2 (0.34) [0.781 to 109] | NA [NA to NA] — There are only two concentration results available for Placebo Patients specified in the listing: Day 85 - 0,658 - below LLOQ Day 89 - 5.93 - above LLOQ
  Week 16 | 27.2 (0.33) [0.369 to 82.7] | NA [NA to NA] — Not calculable because below the lower limit of quantification
  Week 20 | 9.32 (0.35) [0.527 to 36.9] | NA [NA to NA] — Not calculable because below the lower limit of quantification
  Week 24 | 3.66 [0.000 to 18.0] | NA [NA to NA] — Not calculable because below the lower limit of quantification

11. Secondary Outcome: Immunogenicity
Description: Incidence of anti-drug antibodies (ADA) to tralokinumab in serum.
Time Frame: Pre-dose sampling at baseline, Week 8, 12, 16, and 24.
Population: The safety analysis set consist of all randomised participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Tralokinumab | Placebo
Number analyzed (Participants) | 55 | 55
participants
  pre-dose at baseline | 0 (0.31) [0.000 to 0.000] | 1
  Week 8 | 0 (0.29) [12.2 to 92.2] | 1
  Week 12 | 0 (0.34) [5.83 to 116] | 1
  Week 16 | 0 (0.34) [0.781 to 109] | 1
  Week 24 | 0 (0.33) [0.369 to 82.7] | 0

ADVERSE EVENTS:
Time Frame: 24 Weeks
Groups:
- Tralokinumab 300 mg: Tralokinumab 300 mg was administered during study as two subcutaneous 150 mg injections every 2 weeks for 12 weeks starting from Visit 2.
Arm/Group | Placebo | Tralokinumab 300 mg
Serious Adverse Events (participants affected / at risk) | 6/55 | 7/55
Other Adverse Events (participants affected / at risk) | 35/55 | 36/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=55) | Tralokinumab 300 mg (N=55)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 1 (2)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 5 (6) | 5 (5)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 (1) | 0 (0)
SERUM SICKNESS (Immune system disorders) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=55) | Tralokinumab 300 mg (N=55)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
ABDOMINAL PAIN (Gastrointestinal disorders) | 6 (9) | 7 (13)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 10 (12) | 11 (13)
HAEMORRHOIDS (Gastrointestinal disorders) | 1 (1) | 3 (3)
TOOTHACHE (Gastrointestinal disorders) | 1 (1) | 3 (3)
ASTHENIA (General disorders) | 5 (6) | 5 (5)
FATIGUE (General disorders) | 2 (2) | 3 (3)
INJECTION SITE ERYTHEMA (General disorders) | 0 (0) | 3 (10)
INJECTION SITE REACTION (General disorders) | 0 (0) | 3 (3)
PYREXIA (General disorders) | 4 (4) | 6 (7)
INFLUENZA (Infections and infestations) | 4 (5) | 2 (2)
NASOPHARYNGITIS (Infections and infestations) | 5 (6) | 3 (3)
WEIGHT DECREASED (Investigations) | 0 (0) | 3 (3)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (3)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 (5) | 3 (5)
HEADACHE (Nervous system disorders) | 12 (22) | 10 (35)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5)
ALOPECIA (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (4)
TACHYCARDIA (Cardiac disorders) | 2 (2) | 2 (2)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 2 (2)
ABDOMINAL TENDERNESS (Gastrointestinal disorders) | 1 (1) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 2 (2)
DYSPEPSIA (Gastrointestinal disorders) | 2 (2) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 2 (2) | 2 (10)
VOMITING (Gastrointestinal disorders) | 2 (2) | 2 (3)
INFLUENZA LIKE ILLNESS (General disorders) | 2 (3) | 0 (0)
PHARYNGITIS (Infections and infestations) | 2 (3) | 2 (2)
SINUSITIS (Infections and infestations) | 2 (2) | 1 (1)
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
DIZZINESS (Nervous system disorders) | 2 (2) | 2 (2)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less